CLINICAL TRIAL: NCT00624832
Title: A Randomized, Double-blind, Placebo-controlled Study to Demonstrate the Efficacy of Xolair in an Allergen Bronchoprovocation Study in Asthmatic Populations Defined by Serum IgE Concentrations
Brief Title: A Study of Efficacy of New Doses of Xolair to Protect From Allergen Challenge in Groups of Asthma Patients Defined by IgE Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Genentech, Inc. (Industry); Tanox (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIGE025A2210
Record Dates: First submitted 2008-02-18; First posted 2008-02-27 (Estimated); Results first posted 2011-02-14 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Asthma
Keywords: Asthma; allergen challenge; bronchoprovocation; Methacholine challenge; serum Immunoglobulin E; Nitric Oxide; skin prick test
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Xolair (Immunoglobulin E (IgE) = 30-300 IU/mL) (Experimental): Patients with screening Immunoglobulin E (IgE) levels = 30-300 IU/mL. Participants received subcutaneous injections of Xolair (Omalizumab) every 2 weeks or every 4 weeks; dosage dependent on IgE level and body weight.
  Interventions: Drug: Xolair
- Xolair (Immunoglobulin E (IgE) = 700-2000 IU/mL) (Experimental): Patients with screening Immunoglobulin E (IgE) levels = 700- 2000 IU/mL. Participants received subcutaneous injections of Xolair (Omalizumab) every 2 weeks; dosage dependent on IgE level and body weight.
  Interventions: Drug: Xolair
- Xolair (Immunoglobulin E (IgE) = 301-699 IU/mL) (Experimental): Patients with screening Immunoglobulin E (IgE) levels = 301- 699 IU/mL. Participants received subcutaneous injections of Xolair (Omalizumab) every 2 weeks; dosage dependent on IgE level and body weight.
  Interventions: Drug: Xolair
- Placebo (Placebo Comparator): By subcutaneous injection of a solution with a concentration of 125 mg/mL placebo in a supine position: Patients in Xolair (Immunoglobulin E (IgE) = 30-300 IU/mL) group received doses of 150 mg to 375 mg of placebo every 2 or 4 weeks for 12 or 14 weeks. Patients in Xolair (Immunoglobulin E (IgE) = 700- 2000 IU/mL) group received doses of 450 mg, 525 mg, or 600 mg of placebo every 2 weeks for 14 weeks. Patients in Xolair (Immunoglobulin E (IgE) = 301- 699 IU/mL) group received doses of 225 mg to 375 mg of placebo every 2 weeks for 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xolair — Xolair (Omalizumab) dose: 2 x 450 mg, 2 x 525 mg or 2 x 600 mg; subcutaneous injection;
  Arms: Xolair (Immunoglobulin E (IgE) = 30-300 IU/mL); Xolair (Immunoglobulin E (IgE) = 301-699 IU/mL); Xolair (Immunoglobulin E (IgE) = 700-2000 IU/mL)
Drug: Placebo — Matching placebo of Xolair (omalizumab), by subcutaneous injection of a solution with a concentration of 125 mg/mL in a supine position.
  Arms: Placebo

SUMMARY:
This study was intended to demonstrate that patients with standard and high immunoglobulin E (IgE) levels can be protected from allergen induced broncho-constriction by Xolair

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patients, body weight between 40-150 kg aged 18-65 years (inclusive)
* Patients diagnosed with asthma with Forced Expiratory Volume (FEV1) ≥65% of the predicted normal value for the patient
* Positive skin prick test to a specific allergen
* Patients had to demonstrate a Provocative Dose 20% FEV1 decline (PD20) response to an aeroallergen in the graded allergen bronchoprovocation testing (ABP) at screening

Exclusion Criteria:

* Current active smokers
* Patients who have been hospitalized or had emergency treatment for an asthma attack in the 12 months prior to study start
* History of bleeding disorders
* History of drug allergy
* Pregnant women or nursing mothers
* Females of childbearing potential, regardless of whether or not sexually active, if they are not using a reliable form of contraception (surgical contraception or double barrier methods (to be continued for at least two months following last dose) are acceptable).
* Sexually active males who have not been sterilized and are not using a condom
* History of immunocompromise, including a positive HIV
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
* History of drug or alcohol abuse within 12 months of study start

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis investigator site
Locations (6):
- Germany (3):
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Frankfurt
  - Novartis Investigator Site, Munich
- Novartis Investigator Site, Groningen, Netherlands
- South Africa (2):
  - Novartis Investigator Site, Bloemfontein
  - Novartis Investigator Site, Durban

RESULTS

PARTICIPANT FLOW:
Groups:
- Xolair (Immunoglobulin E (IgE) = 700- 2000 IU/mL): Patients with screening Immunoglobulin E (IgE) levels = 700- 2000 IU/mL. Participants received subcutaneous injections of Xolair (Omalizumab) every 2 weeks; dosage dependent on IgE level and body weight.
- Xolair (Immunoglobulin E (IgE) = 301- 699 IU/mL): Patients with screening Immunoglobulin E (IgE) levels = 301- 699 IU/mL. Participants received subcutaneous injections of Xolair (Omalizumab) every 2 weeks; dosage dependent on IgE level and body weight.
- Placebo Comparator: By subcutaneous injection of a solution with a concentration of 125 mg/mL placebo in a supine position: Patients in Xolair (Immunoglobulin E (IgE) = 30-300 IU/mL) group received doses of 150 mg to 375 mg of placebo every 2 or 4 weeks for 12 or 14 weeks. Patients in Xolair (Immunoglobulin E (IgE) = 700- 2000 IU/mL) group received doses of 450 mg, 525 mg, or 600 mg of placebo every 2 weeks for 14 weeks. Patients in Xolair (Immunoglobulin E (IgE) = 301- 699 IU/mL) group received doses of 225 mg to 375 mg of placebo every 2 weeks for 6 weeks.
Period: Overall Study
Arm/Group | Xolair (Immunoglobulin E (IgE) = 30-300 IU/mL) | Xolair (Immunoglobulin E (IgE) = 700- 2000 IU/mL) | Xolair (Immunoglobulin E (IgE) = 301- 699 IU/mL) | Placebo Comparator
Started | 18 | 16 | 10 | 16
Completed | 16 | 15 | 10 | 15
Not Completed | 2 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 1
Not completed — Abnormal Laboratory Value | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Xolair (Immunoglobulin E (IgE) = 30-300 IU/mL) | Xolair (Immunoglobulin E (IgE) = 700- 2000 IU/mL) | Xolair (Immunoglobulin E (IgE) = 301- 699 IU/mL) | Placebo Comparator | Total
Number analyzed (Participants) | 18 | 16 | 10 | 16 | 60
Age Continuous [Mean (Standard Deviation); unit: years] | 36 (11.9) | 29 (11.0) | 26 (6.0) | 34 (10.4) | 32 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 4 | 7 | 26
  Male | 13 | 6 | 6 | 9 | 34

OUTCOME MEASURES:

1. Primary Outcome: Early Phase Allergic Response After Treatment With Study Drug in Active and Placebo Patients
Description: The EAR was defined as the maximum percent drop in forced expiratory volume in one second (FEV1) in the first 30 minutes after the challenge:
  EAR = 100* [ FEV1 (0) - Minimum FEV1 (10, 15, 30 min)] / FEV1 (0). For FEV1 (0), the "best post saline (Control) FEV1" was used. The EAR was analyzed using a linear (ANCOVA) model with a fixed effect for treatment groups and the EAR from the baseline challenge was used as a covariate.
Time Frame: Week 8, Week 16
Population: Safety and Pharmacodynamic (PD) population. Although all patients had baseline EAR not all of them had a value determined for week 8 and 16 reducing the number evaluable for analysis particularly at week 8. Patients of first 2 Xolair groups received placebo treatment were pooled in one placebo group for analysis. No analysis on third Xolair groups.
Measure: Least Squares Mean (Standard Error); unit: Percentage of EAR
Arm/Group | Xolair (Immunoglobulin E (IgE) = 30-300 IU/mL) | Xolair (Immunoglobulin E (IgE) = 700- 2000 IU/mL) | Placebo Comparator
Number analyzed (Participants) | 18 | 16 | 16
Percentage of EAR
  Week 8 (n=12, 12, 13) | 9.3 (3.97) | 5.6 (2.07) | 23.1 (3.57)
  Week 16 (n=14, 15, 15) | 11.8 (3.81) | 5.1 (2.02) | 20.0 (2.43)

2. Secondary Outcome: Late Phase Allergic Response After Treatment With Study Drug in Active and Placebo Patients
Description: Late-phase allergic response (LAR) was only determined for those patients who had an LAR >= 15% at baseline allergen bronchoprovocation testing. For Forced Expiratory Volume, FEV1 (0), the "best post saline (Control) FEV1" was used. LAR (%) = 100*[FEV1 (0) - Minimum FEV1 (3-8h)]/FEV1 (0).
Time Frame: Week 0, Week 8 and Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of LAR
Arm/Group | Xolair (Immunoglobulin E (IgE) = 30-300 IU/mL) | Xolair (Immunoglobulin E (IgE) = 700- 2000 IU/mL) | Placebo Comparator
Number analyzed (Participants) | 18 | 16 | 16
Percentage of LAR
  Week 0 (n=8, 3, 5) | 22.5 (6.12) | 25.7 (12.62) | 27.4 (7.27)
  Week 8 (n=6, 1, 3) | 5.3 (12.13) | -3.5 (0.0) | 19.1 (13.42)
  Week 16 (n=7, 2, 4) | 0.23 (7.109) | 1.5 (1.53) | 12.3 (7.09)

ADVERSE EVENTS:
Time Frame: 18- 26 weeks. Patients were dosed for 6 - 14 weeks depending on treatment group and adverse event data was collected until final study completion evaluation 12 weeks following last dose.
Groups:
- Xolair (IgE= 30- 300 IU/mL): Patients with screening IgE levels= 30-300 IU/mL. Participants received subcutaneous injections of Xolair(Omalizumab) every 2 weeks or every 4 weeks; dosage dependent on IgE level and body weight.
- Xolair (IgE= 700- 2000 IU/mL): Patients with screening IgE levels= 700- 2000 IU/mL. Participants received subcutaneous injections of Xolair(Omalizumab) every 2 weeks; dosage dependent on IgE level and body weight.
- Xolair (IgE= 301- 699 IU/mL): Patients with screening IgE levels= 301- 699 IU/mL. Participants received subcutaneous injections of Xolair(Omalizumab) every 2 weeks; dosage dependent on IgE level and body weight.
- Placebo Comparator: Placebo comparator
Arm/Group | Xolair (IgE= 30- 300 IU/mL) | Xolair (IgE= 700- 2000 IU/mL) | Xolair (IgE= 301- 699 IU/mL) | Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 1/18 | 1/16 | 0/10 | 0/16
Other Adverse Events (participants affected / at risk) | 9/18 | 15/16 | 6/10 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xolair (IgE= 30- 300 IU/mL) (N=18) | Xolair (IgE= 700- 2000 IU/mL) (N=16) | Xolair (IgE= 301- 699 IU/mL) (N=10) | Placebo Comparator (N=16)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Xolair (IgE= 30- 300 IU/mL) (N=18) | Xolair (IgE= 700- 2000 IU/mL) (N=16) | Xolair (IgE= 301- 699 IU/mL) (N=10) | Placebo Comparator (N=16)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 1 | 2
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 2 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 2
Infusion site erythema (General disorders) | 1 | 2 | 0 | 0
Infusion site haematoma (General disorders) | 0 | 1 | 0 | 0
Infusion site induration (General disorders) | 0 | 1 | 0 | 0
Infusion site irritation (General disorders) | 0 | 0 | 1 | 0
Infusion site swelling (General disorders) | 0 | 1 | 0 | 0
Infusion site warmth (General disorders) | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 0 | 1
Injection site swelling (General disorders) | 1 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Eczema infected (Infections and infestations) | 0 | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 1 | 1 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 5 | 1 | 4
Oral herpes (Infections and infestations) | 0 | 2 | 0 | 1
Oral infection (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Pilonidal cyst (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2
Tinea pedis (Infections and infestations) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tooth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood pressure diastolic increased (Investigations) | 0 | 0 | 0 | 1
Blood pressure systolic increased (Investigations) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myosclerosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 5 | 1 | 3
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermographism (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.